CLINICAL TRIAL: NCT00904410
Title: Early Assessment of the Response to Neo-adjuvant Chemotherapy in Breast Cancer Patients With FDG-PET
Acronym: CHIMTEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHIMTEP 0402
Record Dates: First submitted 2007-03-15; First posted 2009-05-19 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: adenocarcinoma; breast
MeSH Terms: conditions — Breast Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: FDG-PET

INTERVENTIONS:
Other: FDG-PET — 370 MBq of FDG one hour before imaging acquisition PET just before neo-adjuvant chemotherapy and just before the second cycle

SUMMARY:
18F-FDG PET, a whole-body imaging technology based on glucose metabolism, can effectively detect subclinical and clinical therapeutic responses at stages that are earlier than those detected by conventional approaches.

We propose to conduct a prospective study to evaluate early therapeutic response using 18F-FDG PET before and after the 1st cycle of neo-adjuvant chemotherapy for breast cancer patients.

Variation of 18F-FDG PET uptake is compared to clinical and echographical tumor response evaluated after 3 cycles of chemotherapy.

The purpose is to estimate the capacity of 18F-FDG PET to differentiate responder and non-responder patients.

DETAILED DESCRIPTION:
Further study details as provided by Centre Oscar Lambret

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Breast cancer treated by neo-adjuvant chemotherapy (T>2cm)
* Measurable lesions ,assessed clinically and by ultrasound
* Delay minimum between biopsy and PET: 15 days
* PS-WHO: 0

Exclusion Criteria:

* T<2cm
* Inflammatory breast cancer (T4d)
* Diabetic patients unbalanced (glycemia>1.40)
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2005-05; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Variation rate of SUV(BSA max)before and after the 1st cycle of neoadjuvant chemotherapy | before and 3 weeks after 1st cycle

SECONDARY OUTCOMES:
Comparison to clinical and ultrasound assessment after the 3rd cycle of chemotherapy | 3 weeks after the 3rd cycle

CONTACTS AND LOCATIONS:
Overall Officials: GAUTHIER Helene, Study Chair — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France